CLINICAL TRIAL: NCT02135224
Title: The Effects of Fentanyl Added to Ropivacaine for Labour Epidural Analgesia on the Progress, Duration or Mode of Delivery: a Randomized, Double Blind Study.
Brief Title: the Effects of Epidural Fentanyl on Vaginal Delivery
Acronym: EFVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Staikou Chryssoula, Assistant Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: M79
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Cervical Dilatation; Bishop Score; Duration of Delivery
MeSH Terms: interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fentanyl (Active Comparator): 20 microgram per hour
  Interventions: Drug: Fentanyl
- Normal saline (Placebo Comparator): 0.4 ml per hour
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Fentanyl
  Arms: Fentanyl
Drug: Normal saline
  Arms: Normal saline

SUMMARY:
The study hypothesis was that epidural fentanyl may accelerate the dilation of the cervix and possibly result in a shorter duration of vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists physical status I or II
* nulliparous
* normal singleton uncomplicated pregnancies of more than 38 weeks
* cephalic presentation of the fetus
* anticipated vaginal delivery
* active stage of labour
* cervical dilatation between 3-5 cm
* regular uterine contractions
* normal cardiotocographic recordings.

Exclusion Criteria:

* medical problems during pregnancy
* BMI≥40 kg m-2
* opioid allergy
* prior administration of opioids or other analgesics

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
cervical dilatation | every 60 min starting from the first epidural dose up to cervical dilatation of 10 cm

SECONDARY OUTCOMES:
Bishop score based on Cervical Position, Effacement, Dilation, Softness and Fetal Station. | every 60 min from the time the first epidural dose is administered up to delivery
  Bishop score is a pre-labor scoring system which reflects the stage of the procedure (mainly the cervix condition) assessing the following: Cervical Position, Effacement, Dilation, Softness and also Fetal Station.

OTHER OUTCOMES:
duration of delivery | min between first epidural dose and delivery of the baby

CONTACTS AND LOCATIONS:
Overall Officials: Chryssoula Staikou, PhD, Principal Investigator — University of Athens
Locations (1):
- Aretaieio Hospital, University of Athens, Athens, Attica, Greece